CLINICAL TRIAL: NCT02807753
Title: Evaluation of Joint Arthropathy Using Ultrasound Technique in Children With Severe Hemophilia Undergoing Prophylaxis Regimen
Brief Title: The Hemophilia Ultrasound Project
Acronym: HUP
Status: Terminated | Type: Observational
Why Stopped: Sponsor funding ended
Sponsor: University of Miami (Other)
Collaborators: Shire (Industry)
Responsible Party: Principal Investigator, Fernando F. Corrales-Medina, MD, University of Miami
Other Study IDs: 20151156
Record Dates: First submitted 2016-06-01; First posted 2016-06-21 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Hemophilia A; Hemophilia B
Keywords: Hemophilia; Arthropathy; Pediatric
MeSH Terms: conditions — Hemophilia A; Hemophilia B; Joint Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Severe Hemophilia A or B: Medical history, physical exam, vital signs,physical therapist targeted exam and ultrasound joint assessment (ankles and knees) every 6 months.
  MRI joint assessment (knees and ankles) at End of Trial Visit (Month 60).
  Interventions: Other: Ankle and Knee Ultrasound Joint Assessment; Other: Ankle and Knee Magnetic Resonance Imaging
- Mild/Moderate Hemophilia A or B: Medical history, physical exam, vital signs,physical therapist targeted exam and ultrasound joint assessment (ankles and knees) every year.
  MRI joint assessment (knees and ankles) at End of Trial Visit (Month 60).
  Interventions: Other: Ankle and Knee Ultrasound Joint Assessment; Other: Ankle and Knee Magnetic Resonance Imaging

INTERVENTIONS:
Other: Ankle and Knee Ultrasound Joint Assessment — Ultrasound Examination of the ankles and knees
Other: Ankle and Knee Magnetic Resonance Imaging — Ankle and Knee Magnetic Resonance Imaging

SUMMARY:
To evaluate the prevalence of subclinical arthropathy in children with severe hemophilia undergoing a prophylaxis regimen and without evidence of target joints, using a validated ultrasound scoring method.

DETAILED DESCRIPTION:
Persons with Hemophilia (A or B) often experience recurrent joint bleeds, most commonly affecting the ankles, knees and elbows. These bleeds can lead to significant pain and disability over time. If recurrent joint bleeds are not managed with prompt and adequate infusions of factor concentrate, the damage caused by the presence of blood in the joint space will eventually result in a condition called debilitating chronic hemophilic arthropathy.

The initiation of and adherence to a prophylactic infusion regimen, starting with the first or second joint bleed, is essential for prevention of progression to arthropathy.

Studies have demonstrated that prophylaxis with recombinant or plasma-derived factor VIII or IX concentrates is effective in preventing clinical joint bleeds and the progression to debilitating joint disease in patients with severe hemophilia A or B respectively. However, for patients on prophylaxis, the absence of symptomatic joint bleeds and/or structural and functional abnormalities of joints on physical examination and plain radiographic images can lead to the erroneous assumption that the prophylaxis is completely effective. It has been established that patients with severe hemophilia are still at risk for subclinical bleeding ("microbleeds") despite seemingly adequate prophylaxis.

Young adults, despite a lifetime on prophylaxis and apparently normal joints are developing arthropathy in their 20's and 30's. Prophylaxis as currently practiced may only be delaying the onset of clinical joint disease.

The recent advancements in ultrasound imaging (US) have been proven to be effective in confirming a joint bleed, monitoring the evolution of a joint bleed and assessing the resolution or recurrence of a bleed. Previous studies have evaluated the prevalence of subclinical arthropathy in young hemophilic adults using both US and MRI techniques and concluded that US is as effective and sensitive as MRI identifying these subclinical joint abnormalities.

However, to the investigators' knowledge, no prior studies have used US technique over an extended period of time to monitor the natural evolution of joint arthropathy in children with hemophilia who are adherent to an established prophylaxis regimen and have no evidence of clinical joint compromise.

The seminal Joint Outcome Study, which confirmed the role of prophylaxis in preventing overt clinical joint disease, mandated a trough residual factor VIII level of 1%. While this trough level significantly decreased overt hemarthroses and joint damage, the evidence suggestive of microbleeds raised a question as to the protection afforded by such a low trough level. Intuitively it would seem as if a higher trough level should confer greater protection against microbleeds, and result in more sustainable joint health. The "ideal" protective trough, has not been established.

The investigators' hypothesis is that US is a valuable imaging technique to monitor the natural evolution of hemophilic arthropathy in children with severe hemophilia A or B who are undergoing prophylaxis regimen and do not manifest clinical evidence of hemophilic arthropathy.

Through this observational study, the investigators will provide valuable information in regards the prevalence, progression and severity of joint abnormalities. The use of US to detect microbleeds before the cumulative damaging effects demonstrable by MRI, will also allow tailoring of treatment and the implementation of new prophylaxis strategies.

ELIGIBILITY:
Inclusion Criteria:

* Severe Hemophilia Cohort:Patients from 0 up to 30 months of age with diagnosis of severe hemophilia A or B defined as a factor VIII:C/IX:C of <1% undergoing prophylaxis regimen with any factor VIII or IX concentrate and without evidence (clinical or by history) of target joint disease.
* Mild/moderate Hemophilia Cohort:Patients from 0 up to 30 months of age with diagnosis of mild hemophilia A or B defined as a factor VIII:C/IX:C of 5-50% and those with diagnosis of moderate hemophilia A or B defined a s a factor VIII:C/IX:C of 1-5% without evidence (clinical or by history) of target joint disease and no history of spontaneous joint bleeds.

Exclusion Criteria:

* Patients with concomitant Hepatitis B, Hepatitis C and HIV viral infections (because of a recognized arthritogen effect).
* Present or prior history of anti FVIII or IX inhibitors.
* Known inflammatory joint disease.
* Established target joint.

Max Age: 30 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Mild, Moderate and Severe Hemophilia A & B patients.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2016-09-16 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2020-12-07 (Actual)

PRIMARY OUTCOMES:
Prevalence and natural progression of subclinical arthropathy (joint changes) in children with severe hemophilia undergoing prophylaxis using a validated ultrasound (HEAD-US) protocol. | 5 years
  Two independent readers will describe all the ultrasonography positive joint findings and/or changes on a standardized spreadsheet; they will also rate and score these changes based on the HEAD-US scale providing a final score for each of the evaluated joints (ankles and knees).
Prevalence and natural progression of subclinical arthropathy (joint changes) in children with mild and/or moderate hemophilia using a validated ultrasound (HEAD-US) protocol. | 5 years
  Two independent readers will describe all the ultrasonography positive joint findings and/or changes on a standardized spreadsheet; they will also rate and score these changes based on the HEAD-US scale providing a final score for each of the evaluated joints (ankles and knees).

SECONDARY OUTCOMES:
Characteristics of subclinical joint changes (time of presentation, natural evolution, etc.) between patients with severe hemophilia and those with mild/moderate hemophilia. | 5 years
  The investigators will describe and compare all the ultrasonography joint findings and/or changes on a standardized spreadsheet in between the two cohort of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando F. Corrales-Medina, MD, Principal Investigator — University of Miami
Locations (4):
- United States (4):
  - University of Florida, Gainesville, Florida
  - The University of Miami - Department of Pediatrics, Miami, Florida
  - University of Kentucky, Lexington, Kentucky
  - Tulane, New Orleans, Louisiana

REFERENCES:
- [Background] Berntorp E. Joint outcomes in patients with haemophilia: the importance of adherence to preventive regimens. Haemophilia. 2009 Nov;15(6):1219-27. doi: 10.1111/j.1365-2516.2009.02077.x. Epub 2009 Jul 29. PMID 19659939
- [Background] Manco-Johnson MJ, Abshire TC, Shapiro AD, Riske B, Hacker MR, Kilcoyne R, Ingram JD, Manco-Johnson ML, Funk S, Jacobson L, Valentino LA, Hoots WK, Buchanan GR, DiMichele D, Recht M, Brown D, Leissinger C, Bleak S, Cohen A, Mathew P, Matsunaga A, Medeiros D, Nugent D, Thomas GA, Thompson AA, McRedmond K, Soucie JM, Austin H, Evatt BL. Prophylaxis versus episodic treatment to prevent joint disease in boys with severe hemophilia. N Engl J Med. 2007 Aug 9;357(6):535-44. doi: 10.1056/NEJMoa067659. PMID 17687129
- [Background] Martinoli C, Della Casa Alberighi O, Di Minno G, Graziano E, Molinari AC, Pasta G, Russo G, Santagostino E, Tagliaferri A, Tagliafico A, Morfini M. Development and definition of a simplified scanning procedure and scoring method for Haemophilia Early Arthropathy Detection with Ultrasound (HEAD-US). Thromb Haemost. 2013 Jun;109(6):1170-9. doi: 10.1160/TH12-11-0874. Epub 2013 Apr 4. PMID 23571706
- [Background] Sierra Aisa C, Lucia Cuesta JF, Rubio Martinez A, Fernandez Mosteirin N, Iborra Munoz A, Abio Calvete M, Guillen Gomez M, Moreto Quintana A, Rubio Felix D. Comparison of ultrasound and magnetic resonance imaging for diagnosis and follow-up of joint lesions in patients with haemophilia. Haemophilia. 2014 Jan;20(1):e51-7. doi: 10.1111/hae.12268. Epub 2013 Sep 24. PMID 24112687
- [Background] Di Minno MN, Iervolino S, Soscia E, Tosetto A, Coppola A, Schiavulli M, Marrone E, Ruosi C, Salvatore M, Di Minno G. Magnetic resonance imaging and ultrasound evaluation of "healthy" joints in young subjects with severe haemophilia A. Haemophilia. 2013 May;19(3):e167-73. doi: 10.1111/hae.12107. Epub 2013 Mar 18. PMID 23496145
- [Background] Doria AS. State-of-the-art imaging techniques for the evaluation of haemophilic arthropathy: present and future. Haemophilia. 2010 Jul;16 Suppl 5:107-14. doi: 10.1111/j.1365-2516.2010.02307.x. PMID 20590865
- [Background] Muca-Perja M, Riva S, Grochowska B, Mangiafico L, Mago D, Gringeri A. Ultrasonography of haemophilic arthropathy. Haemophilia. 2012 May;18(3):364-8. doi: 10.1111/j.1365-2516.2011.02672.x. Epub 2011 Oct 17. PMID 21999202